CLINICAL TRIAL: NCT01673399
Title: Oxytocin Antagonist in Patients With Repeated Failure of Implantation. A Prospective Randomized Placebo-controlled Double-blind Study.
Brief Title: Oxytocin Antagonist in Patients With Repeated Failure of Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Jan Palfijn Gent (Other)
Collaborators: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Dr. Decleer Wim, gynecologist, AZ Jan Palfijn Gent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-000278-49
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Implantation Failure
Keywords: repeated implantation failure (RIF); atosiban; pregnancy
MeSH Terms: interventions — atosiban

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atosiban (Active Comparator): Patients receive a bolus injection of 6.75mg atosiban and following an atosibaninfusion at 18mg/u during 3 hours.
  Interventions: Drug: Atosiban
- placebo (Placebo Comparator): Patients receive a placebo bolus injection (NaCl 0.9%)and an infusion of NaCl 0.9% during 3 hours
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Atosiban — Bolus atosiban 6.75mg + infusion atosiban 18mg/u during 3 hours. once administered starting 1 hour before embryotransfer.
  Arms: Atosiban
Drug: placebo
  Arms: placebo

SUMMARY:
In this study the investigators compare the usual way of embryo transfer (without medication) with an embryo transfer while administering oxytocine antagonist. This to improve implantation and increase the pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* IVF/ ICSI patients below 38 years
* 2e to 6e IVF-cycle

Exclusion Criteria:

* patients with endocrinological diseases or problems

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
implantation rate | 16 days from eggretrieval
  the number of patients that show a positive serum blood pregnancy test

SECONDARY OUTCOMES:
pregnancy rate | 12 weeks
  The number of patients with an ongoing first trimester pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Jan Palfijn, Ghent, Oost-vlaanderen, Belgium

REFERENCES:
- [Derived] Craciunas L, Tsampras N, Kollmann M, Raine-Fenning N, Choudhary M. Oxytocin antagonists for assisted reproduction. Cochrane Database Syst Rev. 2021 Sep 1;9(9):CD012375. doi: 10.1002/14651858.CD012375.pub2. PMID 34467530